CLINICAL TRIAL: NCT03490487
Title: Electroclinical Effect of Steroid in Patients With Benign Childhood Epilepsy With Centrotemporal Spikes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khalaf A Sayed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DS
Record Dates: First submitted 2018-02-18; First posted 2018-04-06 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Benign Childhood Epilepsy With Centrotemporal Spikes
MeSH Terms: conditions — Epilepsy, Rolandic | interventions — Carbamazepine; Valproic Acid; Oxcarbazepine; Levetiracetam; Steroids; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A antiepileptic (Active Comparator): will receive conventional antiepileptic drugs only
  Interventions: Drug: conventional antiepileptic drugs
- B steroid (Experimental): will receive oral steroid for 3 months beside conventional antiepileptic drugs
  Interventions: Drug: conventional antiepileptic drugs; Drug: oral steroid

INTERVENTIONS:
Drug: conventional antiepileptic drugs — will receive conventional antiepileptic drugs only. EEG, attention deficit hyperactivity disorder test and intelligence quotient will be done before and 3 months after treatment.
  Other Names: carbamazepine, valproate, oxcarbazepine or levetiracetam
Drug: oral steroid — will receive oral steroid for 3 months beside conventional antiepileptic drugs. EEG, attention deficit hyperactivity disorder test and intelligence quotient will be done before and 3 months after treatment.
  Other Names: Prednisolone
  Arms: B steroid

SUMMARY:
Benign epilepsy with centro-temporal spikes is the most common type of focal epilepsy in children. It is known to be age-dependent and presumably genetic. Age of onset ranges from one to fourteen years and it represents fifteen percent to twenty five percent of epilepsy in children under 15 years of age.

DETAILED DESCRIPTION:
Generally, Benign epilepsy with centro-temporal spikes is characterized by infrequent focal sensorimotor seizures in the face during sleep, which may secondarily generalize, along with spike-wave discharges, reflecting nonlesional cortical excitability from rolandic regions.

The prognosis is usually considered to be excellent. Over the past years, however, some investigators have questioned whether Benign epilepsy with centro-temporal spikes is indeed benign, considering the variety of different presentations associated with the disorder.It is not uncommon for Benign epilepsy with centro-temporal spikes to be associated with neuropsychological deficits, such as linguistic, cognitive, and behavioral impairment. In particular, reading difficulties and speech/language disorders are more common in children with Benign epilepsy with centro-temporal spikes than in healthy controls.Various neuropsychological deficits seem to be very dependent on the spike index, as well as the predominant localization of epileptiform discharges.Furthermore, the frequency of epileptiform discharges is closely related not only to the degree of neuropsychological deficits, but also to an atypical evolution of benign epilepsy with centro-temporal spikes.

The high comorbid prevalence of attention deficit hyperactivity disorder and epilepsy suggests that there is a bidirectional relationship between these disorders .Cognitive impairment and attention problems are particularly crucial issues in children with epilepsy who are in a vigorous phase of neurodevelopment.

Resolution of continuous spike-and-wave during sleep had been achieved with conventional antiepileptic drugs including ethosuximide, valproic acid, levetiracetam, and sulthiame. When these agents fail to normalize the EEG, a trial with second-line agents such as steroids or high-dose diazepam is attempted.

ELIGIBILITY:
Inclusion Criteria:

* History and EEG findings of benign epilepsy with centrotemporal spikes

Exclusion Criteria:

* Genetic disorders.
* Metabolic or neurodegenerative disease.
* Gross motor delay.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
To detect the effect of oral steroids on normalization of sleep EEG. | 3 months
  follow up Electroencephalography and calculation of spike-wave index before and after three months of treatment with steroid.Any reduction in spike wave index on electroencephalograph after receiving steroid will be considered improvement.The EEG technicians will be requested to perform a prolonged daytime nap EEG. The researcher first will look at the full sleep recording and visually pick the epoch with the highest spike density. The counting start with a page of a high spike density and continued for 10 consecutive minutes. Each page will be scored separately. Each second which contained spikes, either focal or generalized, will be considered positive, and the total number of positive seconds per page will be calculated as percents of the whole page. At the end of the counting, an average of 60 pages (10 min) will be performed and then displayed in terms of the nearest ten percentile number.
To detect the effect of oral steroids regarding improvement of cognitive functions of patients with BECTS. | 3 months
  Intelligence quotient assessment with Stanford-Binet scales will be done before and after three months of treatment with steroid. Stanford-Binet Intelligence Scale (Fourth Edition) score: very superior (140 and above), superior (120-139), high average (110-119), normal average (90-109), low average (80-89), borderline defective (70-79), mentally defective (30-69). Higher scores will be considered a better or outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal A Abdelal, MD, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fejerman N, Caraballo R, Tenembaum SN. [Atypical evolutions of benign partial epilepsy of infancy with centro-temporal spikes]. Rev Neurol. 2000 Aug 16-31;31(4):389-96. Spanish. PMID 11008297
- [Background] Ay Y, Gokben S, Serdaroglu G, Polat M, Tosun A, Tekgul H, Solak U, Kesikci H. Neuropsychologic impairment in children with rolandic epilepsy. Pediatr Neurol. 2009 Nov;41(5):359-63. doi: 10.1016/j.pediatrneurol.2009.05.013. PMID 19818938
- [Background] Danielsson J, Petermann F. Cognitive deficits in children with benign rolandic epilepsy of childhood or rolandic discharges: a study of children between 4 and 7 years of age with and without seizures compared with healthy controls. Epilepsy Behav. 2009 Dec;16(4):646-51. doi: 10.1016/j.yebeh.2009.08.012. Epub 2009 Oct 29. PMID 19879197
- [Background] Clarke T, Strug LJ, Murphy PL, Bali B, Carvalho J, Foster S, Tremont G, Gagnon BR, Dorta N, Pal DK. High risk of reading disability and speech sound disorder in rolandic epilepsy families: case-control study. Epilepsia. 2007 Dec;48(12):2258-65. doi: 10.1111/j.1528-1167.2007.01276.x. Epub 2007 Sep 10. PMID 17850323
- [Background] Kanemura H, Sano F, Aoyagi K, Sugita K, Aihara M. Do sequential EEG changes predict atypical clinical features in rolandic epilepsy? Dev Med Child Neurol. 2012 Oct;54(10):912-7. doi: 10.1111/j.1469-8749.2012.04358.x. Epub 2012 Jul 4. PMID 22759211
- [Background] Kwon S, Hwang TG, Lee J, Kim DK, Seo HE. Benign childhood epilepsy with centrotemporal spikes: to treat or not to treat. J Epilepsy Res. 2013 Jun 30;3(1):1-6. doi: 10.14581/jer.13001. eCollection 2013 Jun. PMID 24649464
- [Background] Kwon S, Seo HE, Hwang SK. Cognitive and other neuropsychological profiles in children with newly diagnosed benign rolandic epilepsy. Korean J Pediatr. 2012 Oct;55(10):383-7. doi: 10.3345/kjp.2012.55.10.383. Epub 2012 Oct 29. PMID 23133485
- [Background] Inutsuka M, Kobayashi K, Oka M, Hattori J, Ohtsuka Y. Treatment of epilepsy with electrical status epilepticus during slow sleep and its related disorders. Brain Dev. 2006 Jun;28(5):281-6. doi: 10.1016/j.braindev.2005.09.004. Epub 2006 Jan 10. PMID 16376508
- [Background] Kramer U, Sagi L, Goldberg-Stern H, Zelnik N, Nissenkorn A, Ben-Zeev B. Clinical spectrum and medical treatment of children with electrical status epilepticus in sleep (ESES). Epilepsia. 2009 Jun;50(6):1517-24. doi: 10.1111/j.1528-1167.2008.01891.x. Epub 2008 Nov 19. PMID 19054417
- [Background] Guerrini R, Genton P, Bureau M, Parmeggiani A, Salas-Puig X, Santucci M, Bonanni P, Ambrosetto G, Dravet C. Multilobar polymicrogyria, intractable drop attack seizures, and sleep-related electrical status epilepticus. Neurology. 1998 Aug;51(2):504-12. doi: 10.1212/wnl.51.2.504. PMID 9710026
- [Background] Scheltens-de Boer M. Guidelines for EEG in encephalopathy related to ESES/CSWS in children. Epilepsia. 2009 Aug;50 Suppl 7:13-7. doi: 10.1111/j.1528-1167.2009.02211.x. PMID 19682043
- [Background] Chou IC, Chang YT, Chin ZN, Muo CH, Sung FC, Kuo HT, Tsai CH, Kao CH. Correlation between epilepsy and attention deficit hyperactivity disorder: a population-based cohort study. PLoS One. 2013;8(3):e57926. doi: 10.1371/journal.pone.0057926. Epub 2013 Mar 6. PMID 23483944